CLINICAL TRIAL: NCT07264894
Title: ZSDT for the Treatment of Recurrent Refractory Mantle Cell Lymphoma After BTK Inhibitor Failure: a Multi-center Prospective Clinical Trial
Brief Title: ZSDT for the Treatment of R/R Mantle Cell Lymphoma After BTK Inhibitor Failure: a Multi-center Prospective Clinical Trial
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhengzhou University (Other)
Responsible Party: Principal Investigator, Mingzhi Zhang, Professor, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-KY-0057-004
Record Dates: First submitted 2025-11-16; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Mantle Cell Lymphoma (MCL)
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ZSDT regemin (Experimental): This study enrolled 30 patients with relapsed refractory mantle cell lymphoma (MCL). The treatment protocol included: selinexor 60mg once daily on days 1 and 8, zuberitamab 375 mg/m² on day 0, Dexamethasone 20 mg on days 1-3 and 8-9, and thalidomide 200 mg on days 1-21. Each treatment cycle lasted 21 days, with six consecutive cycles. Patients achieving complete remission (CR) or partial response (PR) would receive a year-long maintenance therapy of zuberitamab 375 mg/m² every three months and selinexor 60 mg daily on days 1 and 8. Patients experiencing disease progression (PD) would be excluded from the study.
  Interventions: Drug: ZSDT regimen

INTERVENTIONS:
Drug: ZSDT regimen — The study is based on the R2 protocol and preclinical and clinical studies of selinexor. For relapsed refractory MCL patients who had received BTK inhibitors: selinexor 60mg once daily on days 1 and 8, zuberitamab 375 mg/m² on day 0, Dexamethasone 20 mg on days 1-3 and 8-9, and thalidomide 200 mg on days 1-21. Each treatment cycle lasted 21 days, with six consecutive cycles. Patients achieving complete remission (CR) or partial response (PR) would receive a year-long maintenance therapy of zuberitamab 375 mg/m² every three months and selinexor 60 mg daily on days 1 and 8. Patients experiencing disease progression (PD) would be excluded from the study.

SUMMARY:
For relapsed/refractory mantle cell lymphoma patients that previously treated with BTK inhibitors: The first part involves 6 cycles of combined therapy with zuberitamab, selinexor, dexamethasone, and thalidomide. This targeted combination regimen can enhance efficacy while reducing toxic side effects. The second part utilizes Zuberitamab plus selinexor for maintenance consolidation therapy, thereby reducing relapse and prolonging survival.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-70, ECOG score 0-2(including ages 18 and 70);
2. Overall Survival > 6 months;
3. The diagnosis of mantle cell lymphoma was confirmed by histopathology. 4.At least one measurable lesion;

5.Acceptable hematologic parameters, no contraindications to chemotherapy, absolute neutrophil ≥1.0 × 10 ^ 9 L, platelet ≥75 × 10 ^ 9 L, hemoglobin ≥80 g/L (except for patients with bone marrow infiltration) 6.Liver function: direct bilirubin ≤1.5 × upper limit , Alanine transaminase or aspartate transaminase ≤2.5 × upper limit , Alkaline phosphatase≤3 × ULN in patients without non-bone involvement 7.Renal function: serum creatinine ≤1.5 ×ULN 5; 8.Women of Childbearing Potential (WOBCP) or men and their WOBCP partners should agree to take effective contraceptive measures from the signing of ICF and WOBCP must undergo a serum pregnancy test within seven days before the first medication and the results are negative; 9.Recurrent refractory patients after BTK inhibitor treatment; 10.The subjects voluntarily participate the study.

Exclusion Criteria:

1. Refusing to take blood samples;
2. Previous allergies to any of the medications in the regimen;
3. Pregnant and lactating women;
4. The researchers believe that major diseases can cause interference in the trial.;
5. Combined with other tumors.;
6. There are drug-related contraindications to treatment in the protocol;
7. People with severe mental illness;
8. Participating in other clinical trials;
9. Other serious diseases that may limit the subject's participation in this trial, such as: uncontrolled diabetes mellitus; Severe cardiac insufficiency (NYHA classification II or above); Acute coronary syndrome within the past 6 months; Coronary revascularization such as stenting, coronary artery bypass surgery, and other heart and large vessel related surgeries in the past 6 months; Severe arrhythmias include frequent premature ventricular episodes, ventricular tachycardia, rapid atrial fibrillation/atrial flutter, and severe bradycardia. Uncontrolled hypertension: systolic blood pressure > 150 mmHg, diastolic blood pressure > 100 mmHg. Gastric ulcer (gastric ulcer judged by the investigator to be at risk of perforation); Active autoimmune disease (e.g., systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjögren's syndrome, autoimmune thrombocytopenia, etc.); Severe respiratory diseases (such as obstructive pulmonary disease and history of bronchospasm), etc.;
10. In the opinion of the investigators, it is not suitable for enrollment;
11. Hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer test is not within the normal reference value; Those who are positive for hepatitis C virus (HCV) antibody and positive for hepatitis C virus (HCV) RNA in peripheral blood; Those who are positive for human immunodeficiency virus (HIV) antibodies; Those who test positive for syphilis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
CRR | From enrollment to the end of treatment at 8 weeks
  comple remission rate

CONTACTS AND LOCATIONS:
Overall Officials: Professor Zhang, Principal Investigator — The first affliated hospital of ZhengZhou University
Locations (1):
- The first affiliated hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No